CLINICAL TRIAL: NCT03876106
Title: A Phase 1, Open-Label, Dose Escalation Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy Study of Topically Administered LUT014 in Metastatic Colorectal Cancer Patients With EGFR Inhibitor Induced Acneiform Lesions
Brief Title: A Study of LUT014 in Patients With Metastatic Colorectal Cancer With EGFR Inhibitor Induced Acneiform Lesions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lutris Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: L-01-01
Record Dates: First submitted 2019-03-11; First posted 2019-03-15 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: EGFR Inhibitor Induced Acneiform Lesions
MeSH Terms: interventions — LUT014

STUDY DESIGN:
Intervention Model Description: 3+3 Dose escalation of LUT014
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LUT014 dose level 1 (Experimental): LUT014 will be topically applied to the face, neck, and upper portion of the anterior and posterior chest once a day for 4 weeks.
  Interventions: Drug: LUT014
- LUT014 dose level 2 (Experimental): LUT014 will be topically applied to the face, neck, and upper portion of the anterior and posterior chest once a day for 4 weeks.
  Interventions: Drug: LUT014
- LUT014 dose level 3 (Experimental): LUT014 will be topically applied to the face, neck, and upper portion of the anterior and posterior chest once a day for 4 weeks.
  Interventions: Drug: LUT014

INTERVENTIONS:
Drug: LUT014 — Topical

SUMMARY:
The purpose of this phase 1, multicenter study is to evaluate the safety, tolerability and preliminary efficacy of LUT014 in adult metastatic colorectal cancer patients with EGFR Inhibitor induced acneiform lesions

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mCRC;
* Currently being treated with an FDA approved EGFRI for the treatment of mCRC, including but not limited to Erbitux® (cetuximab) Injection and Vectibix® (panitumumab) Injection, as directed by the approved labeling;
* Treatment with the FDA approved EGFRI initiated within 12 weeks prior to the Screening Visit;
* Grade 1 or 2 acneiform lesions at the Screening and Baseline (Day 0) Visits; A minimum of 3 subjects per dose cohort must have Grade 2 non-infected acneiform lesions at the Screening and Baseline (Day 0) Visits;
* Age ≥18 years at the time of signing the informed consent form (ICF);
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2;
* Expected life expectancy greater than 3 months;
* Subject can understand and sign the ICF, can communicate with the Investigator, can understand and comply with the requirements of the protocol, and can apply the study drug by himself/herself or has a care giver that can apply the drug;
* Women of childbearing potential (WCBP) must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at baseline (Day 0);
* WCBP must agree to abstain from sex or use an adequate method of contraception from the time of informed consent through the Day 55 Visit and for 90 days after the last dose of study drug (LUT014);
* Males must abstain from sex with WCBP or use an adequate method of contraception from the time of informed consent through the Day 55 Visit and for 90 days after the last dose of study drug (LUT014).

Exclusion Criteria:

* Active infection;
* Significant skin disease other than EGFRI induced acneiform lesions;
* Any cancer other than mCRC within 3 years of Screening;
* Any condition which, in the opinion of the Investigator, places the subject at unacceptable risk if he/she were to participate in the study;
* Clinically relevant serious co-morbid medical conditions including, but not limited to, unstable angina, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled cardiac arrhythmias, chronic obstructive or chronic restrictive pulmonary disease, active central nervous system (CNS) disease uncontrolled by standard of care, known positive status for human immunodeficiency virus (HIV) and/or active hepatitis B or C, cirrhosis, or psychiatric illness/social situations that would limit compliance with study requirements;
* Pregnant or lactating;
* Treatment with an EGFRI other than those specified in the inclusion criteria within 30 days or 5 half-lives of the drug prior to Screening, whichever is longer;
* Treatment with a serine/threonine-protein kinase B-Raf (B-Raf) inhibitor, including but not limited to Zelboraf® (vemurafenib), Tafinlar® (dabrafenib), BraftoviTM (encorafenib), and Nexavar® (sorafenib), within 30 days or 5 half-lives of the drug prior to Screening, whichever is longer;
* Treatment with a systemic antibiotic within 7 days prior to Screening;
* Treatment with a topical corticosteroid to the face, neck, or upper portion of the anterior or posterior chest within 14 days prior to Screening or treatment with a systemic corticosteroid within 14 days prior to Screening, except for low dose systemic corticosteroids (e.g., 8-20 mg dexamethasone or comparable) given for up to one or two days every two weeks as part of standard of care for the prevention or treatment of chemotherapy-induced nausea and vomiting (CINV) for subjects being treated with FDA-approved EGFRI and chemotherapy combinations for mCRC;
* Treatment with an oral retinoid within 7 days prior to Screening;
* Treatment with another investigational drug within 30 days or 5 half-lives of drug prior to Screening, whichever is longer;
* Known hypersensitivity to the inactive ingredients of the study drug (LUT014).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (maximum tolerated dose, MTD) of LUT014 topically applied qd for 4 weeks in metastatic colorectal cancer (mCRC) patients with epidermal growth factor receptor inhibitor (EGFRI) induced acneiform lesions. | From Day 0 (following administration of the first dose of study drug) through the Day 55

SECONDARY OUTCOMES:
Maximum concentration (Cmax) in plasma after a single administration and after qd administrations for 8 days | Pre-dose through Day 8
Time to maximum concentration (Tmax) in plasma after a single administration and after qd administrations for 8 days | Pre-dose through Day 8
Area under the concentration-time curve from time zero to last measurable concentration (AUC0-T) | Pre-dose through Day 8
Area under the concentration-time cure from time zero extrapolated to infinity (AUC0-∞) | Pre-dose through Day 8
Plasma elimination half-life (t1/2) | Pre-dose through Day 8
Plasma clearance (CL) | Pre-dose through Day 8
Volume of distribution (Vd) | Pre-dose through Day 8
NCI, Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 skin and subcutaneous tissue disorders grading scale performed locally by the Investigator | Pre-dose through Day 55
  The scale contains 5 grades from 1 which demonstrates the mild form of the disease up to 5, defined as death.
MASCC Study Group EGFRI-dermatologic AE grading by central reader based on photographs | Pre-dose through Day 55
Functional Assessment of Cancer Therapy-EGFRI 18 (FACT-EGFRI-18) on health-related quality of life (HRQoL) questionnaire | Pre-dose through Day 55
  FACT-EGFRI-18 is a patient-reported outcomes questionnaire developed to assess the effect of EGFRI on health-related quality of life The questionnaire includes 18 questions, each should be graded from 0, not suffering from this side effect at all, up to 4, suffering greatly from this side effect

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - UCLA Health Santa Monica - Cancer Care, Los Angeles, California
  - Washington University School of Medicine-Dermatology, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan